CLINICAL TRIAL: NCT02602184
Title: Prospective, Placebo-controlled, Double Blind, Randomized Intra-individual Comparative Clinical Study to Assess the Safety and Efficacy of AR/101 Compared to Placebo in Accelerating Re-epithelialization of Split Thickness Wounds
Brief Title: Safety and Efficacy of AR/101 in Accelerating Re-epithelialization of Split Thickness Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arava Bio Tech Ltd. (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NU-AR-2015-01
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-11

CONDITIONS: Wounds and Injuries
Keywords: skin regeneration; re-epithelialization; split thickness wounds; Abdominoplasty
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR/101 (Experimental): Topically treatment with AR/101+Standard of Care once daily for up to 21 days. Daily treatment will include application of AR/101 drug to the wound and coverage with dressing (SoC). Subjects who are scheduled for an elective abdominoplasty at the practice of the principal investigator will have superficial split thickness wounds created on their abdomen according to protocol about 4 weeks prior to their scheduled abdominoplasty. A total of 8 split thickness (5X5 cm, 0.0254 mm in thickness) wounds will be distributed on the abdomen between the umbilicus and the suprapubic hairline. 4 of the wounds will be treated with AR/101.
  Interventions: Drug: AR/101
- Placebo (Placebo Comparator): Topically treatment with Placebo + Standard of Care once daily for up to 21 days. Daily treatment will include application of placebo control to the wound and coverage with dressing (SoC). Subjects who are scheduled for an elective abdominoplasty at the practice of the principal investigator will have superficial split thickness wounds created on their abdomen according to protocol about 4 weeks prior to their scheduled abdominoplasty. A total of 8 split thickness (5X5 cm, 0.0254 mm in thickness) wounds will be distributed on the abdomen between the umbilicus and the suprapubic hairline. 4 of the wounds will be treated with Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR/101
  Arms: AR/101
Drug: Placebo
  Arms: Placebo

SUMMARY:
This clinical study will be a prospective, placebo-controlled, double-blind, randomized and centrally evaluated intra-individual comparative study to assess the safety and efficacy of AR/101 concomitantly administered with Standard of Care (SoC) in accelerating re epithelialization of split thickness wounds compared with placebo and concomitantly with SoC, in the pannus of volunteers undergoing elective abdominoplasty.

DETAILED DESCRIPTION:
This clinical study will be a prospective, placebo-controlled, double-blind, randomized and centrally evaluated intra-individual comparative study to assess the safety and efficacy of AR/101 concomitantly administered with SoC in accelerating re epithelialization of split thickness wounds compared with placebo and concomitantly with SoC, in the pannus of volunteers undergoing elective abdominoplasty.

Total duration of the treatment in the study is 21 days. The patients will be treated with AR/101 or placebo until complete re epithelialization or up to 21 days, whichever comes first. Evaluation and treatment will be done daily in the outpatient clinic. Throughout the study, safety data on adverse events will be collected.

All patients will receive standard supportive care and dressing supplies concomitantly with AR/101 or placebo.

Volunteers who are scheduled for an elective abdominoplasty at the practice of the principal investigator will have superficial split thickness wounds created on their abdomen according to protocol about 4 weeks prior to their scheduled abdominoplasty. A total of 8 split thickness (5X5 cm, 0.0254 mm in thickness) wounds will be distributed on the abdomen between the umbilicus and the suprapubic hairline. All patients will have to agree to daily treatment in the hospital clinic by professional staff through the study duration. Degree of re-epithelialization will be assessed photographically and confirmed by the absence of drainage on wound dressings.

All treated wounds that achieve complete re-epithelialization within the study period will be evaluated for the retention of an intact epithelium at the end of the study (22 days). At the time of the subject's abdominoplasty surgery, the pannus of each subject will be surgically removed as part of the abdominoplasty procedure, and skin samples will be harvested from the excised pannus for further histologic and molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 25-55 years old
2. Patient has chosen to undergo and scheduled an elective cosmetic abdominoplasty
3. Subject has sufficient excess abdominal tissue to qualify for a standard elective abdominoplasty. [Standard abdominoplasty including minor liposuction of the abdominal flap, mons pubis (female patients), and flanks.]
4. Subject is able to tolerate up to a 4 hour abdominoplasty operation under conscious sedation and local tumescent anesthesia, or general anesthesia.
5. Subject donor site can accommodate up to 8, 5X5 cm split thickness wounds which will be distributed on the abdomen between the umbilicus and the suprapubic hairline as per the Principal Investigator.
6. Subject is medically healthy with normal laboratory and ECG screening results (or with values that are outside of the normal range but not considered clinically significant, as per the Principal Investigator).
7. Subject is ready to comply with all study requirements, including: visiting the trial site for daily dressing changes and photo documentation for 22 days
8. The patient is willing and able to adhere to the protocol regimen.
9. For female subjects only, the subject is either:

1. Surgically sterile. 2. At least 1 year post-menopausal. 3. Subject has consented to using one of the following acceptable methods of birth control for the times specified below:

1. Intra-uterine device (IUD) in place for at least 3 months prior to screening visit and through study completion.
2. Barrier method (condom or diaphragm) for at least 14 days prior to screening through study completion.
3. Spermicide for at least 14 days prior to screening through study completion.
4. Stable hormonal contraceptive for at least 3 months prior to screening visit through study completion.
5. Surgical Sterilization (vasectomy) of partner at least 6 months prior to screening visit through study completion.

   10. Subject is non-smoker or stopped smoking at least 6 weeks before study start; subject has negative cotinine test.

   11. The patient is able to read, understand, and has signed the informed consent form. In case of compromised mental capacity, approval and signature of a legal guardian is required.

   Exclusion Criteria:
   1. Subject has prior history of panniculectomy, circumferential lipectomy, lower body lift, belt lipectomy.
   2. Subject has combined procedures (such as concurrent breast augmentation, etc.).
   3. Subject has body mass index (BMI) < 20 or > 35.
   4. Subject has existing scars or significant striae on the abdominal pannus to be removed during the abdominoplasty procedure, with the exception of vertical midline scars or scars at the periphery (such as transverse Caesarian scars at the level of the pubis) that would not interfere with this study.
   5. Subject has a systemic infection or significant local infection such as cellulitis, purulent drainage, gangrene, or necrosis at the target wound site, as well as nonviable tissue, sinus tracts or tunnels that cannot be removed by debridement.
   6. Subject has a skin disorder which is chronic or currently active (e.g. cutis laxa, radiation damage, sun damage, etc.) or other skin condition which in the opinion of the investigator will adversely affect the healing ability of the patient according to the protocol.
   7. Subject has a history of skin sensitivity (dermatitis) to the dressings to be utilized during the course of this study.
   8. Subject has had aggressive liposuction or lipodissolve therapy that resulted in inadequate subcutaneous fat so that the skin in the study area is compromised.
   9. Subject has an abdominal hernia that in the opinion of the investigator would interfere with the conduct of this study.
   10. Subject has previous history or presence of malignancies, or of any illness or condition that may impair re-epithelialization or healing, immune deficiency or connective tissue disease (e.g., SLE, AIDS), neurological disease (e.g., multiple sclerosis), circulatory disease, peripheral vascular disease, dialysis due to renal disease, active hepatic disease, significant cardiovascular, pulmonary, hematological, gastrointestinal, endocrine, immunologic, dermatologic or psychiatric abnormalities.
   11. Subject has a previous medical documentation of positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
   12. Patients with current known history of diabetes
   13. Patient is receiving, or plans to while on study, or has received within 14 days prior to Visit 0 any medication (with exception of hormonal contraceptives and HRT) known to impair re-epithelialization or healing, including but not limited to: steroids (topical, injected, consumed, or inhaled) or other immune modulators, corticosteroids, immuno-suppressive drugs, cytotoxic agents, radiation therapy and chemotherapy, NSAIDs, aspirin or other blood thinners; OR any other treatment that in the investigator's judgment will affect wound healing or bleeding.
   14. Subject has a history or presence of alcoholism or drug abuse within the 2 years prior to Visit 0.
   15. Female patient who is pregnant, or was pregnant during the 12 months prior to inclusion in the study, or nursing, or of childbearing potential which is not using adequate contraception.
   16. Patients who in the opinion of the investigator, for any reason other than those listed above will not be able to complete the study per protocol.
   17. Participation in another clinical trial within 30 days prior to the Screening Visit or during this study.
   18. History of mental illness that would preclude completion of the study
   19. Subject has history of anaphylactic reactions.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The number of days, per wound within a subject, from treatment initiation to complete re epithelialization. | Up to 21 days

SECONDARY OUTCOMES:
The number of days, per wound within a subject, from treatment initiation to reach 50% re-epithelialization | Up to 21 days
The number of days, per wound within a subject, from treatment initiation to reach 75% re-epithelialization | Up to 21 days
Percentage of split thickness wounds with full re-epithelialization | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galiano, MD FACS, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States